CLINICAL TRIAL: NCT06502912
Title: Association Between Iron Reserves and Perioperative Neurocognitive Disorders
Status: Completed | Type: Observational
Sponsor: Chinese PLA General Hospital (Other)
Responsible Party: Principal Investigator, Weidong Mi, Director (Cheif expert of National key research and development program of China 2018YFC2001900), Chinese PLA General Hospital
Other Study IDs: PLAGH-AOC-R02
Record Dates: First submitted 2024-07-02; First posted 2024-07-16 (Actual); Last update posted 2024-07-16 (Actual); Status verified 2024-07

CONDITIONS: Perioperative Neurocognitive Disorders
Keywords: iron reserves; Perioperative neurocognitive disorders; elderly; iron overload
MeSH Terms: conditions — Iron Overload

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- elderly patients (aged ≥ 65 years): elderly patients undergoing non-neurosurgical and non-cardiac procedures
  Interventions: Other: no intervention

INTERVENTIONS:
Other: no intervention — no intervention

SUMMARY:
Iron metabolism disorder have been identified as the pivotal contributor in the pathogenesis and progression of perioperative neurocognitive disorders. However, the association between iron reserves and perioperative neurocognitive disorders risk remains elusive. This retrospective cohort study aimed to explore the impact of preoperative serum ferritin levels on the risk of postoperative delirium in elderly patients undergoing non-neurosurgical and non-cardiac procedures.

ELIGIBILITY:
Inclusion Criteria:

* Geriatric surgical patients ≥65 years old

Exclusion Criteria:

* preoperative use of antipsychotics
* diagnosis or history description of preoperative cognitive disorders including dementia and Parkinson's

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Study Population: hospital based group
Sampling Method: Non-Probability Sample
Enrollment: 12984 (Actual)
Dates: Start 2014-01-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2021-12-31 (Actual)

PRIMARY OUTCOMES:
Number of participants with postoperative delirium | Within the first seven days following surgery
  Medical chart review was used for postoperative delirium determination in this study. The defining criteria were as follows: 1) delirium-related terms included in postoperative medical records or 2) postoperative record of delirium or psychotropic drugs treatment.

CONTACTS AND LOCATIONS:
Overall Officials: Weidong Mi, PhD, Study Chair — Chinese PLA General Hospital

IPD SHARING:
Plan to Share IPD: Undecided